CLINICAL TRIAL: NCT04550715
Title: Optimized Interventions to Prevent Opioid Use Disorder Among Adolescents and Young Adults in the Emergency Department
Brief Title: Prevention Interventions for Opioid Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Maureen A Walton, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00177625; UG3DA050173 (NIH)
Record Dates: First submitted 2020-08-25; First posted 2020-09-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use
Keywords: opioid misuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brief intervention (BI) then Portal (Experimental): The BI will be delivered at intake and the portal will occur for 4 weeks starting at intake.
  Interventions: Behavioral: Brief intervention (BI); Behavioral: Portal
- Brief intervention (BI) then Enhanced Usual Care (EUC) (Experimental): The BI will be delivered at intake and EUC will be added 4 weeks later.
  Interventions: Behavioral: Brief intervention (BI); Behavioral: Enhanced Usual Care (EUC)
- Enhanced Usual Care (EUC) then Portal (Experimental): EUC will be delivered at intake and the portal will occur for 4 weeks starting at intake.
  Interventions: Behavioral: Portal; Behavioral: Enhanced Usual Care (EUC)
- Enhanced Usual Care (EUC) then EUC (Active Comparator): EUC will be delivered at intake and delivered again 4 weeks later.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Brief intervention (BI) — A remote brief intervention delivered by health coaches that uses Motivational Interviewing to address opioid misuse and risk factors. Remote health coaches use a web-based clinician support guide to maintain fidelity, while tailoring the session to unique participant factors.
  Arms: Brief intervention (BI) then Enhanced Usual Care (EUC); Brief intervention (BI) then Portal
Behavioral: Portal — Remote health coaches will push tailored messages to participants over a 4-week period. The messages will use Motivational Interviewing strategies. The messages are designed to elicit a response from the participant. Health coaches will also respond to participant replies consistent with Motivational Interviewing over a course of 4 weeks.
  Arms: Brief intervention (BI) then Portal; Enhanced Usual Care (EUC) then Portal
Behavioral: Enhanced Usual Care (EUC) — The brochure covers educational topics like opioid storage and disposal and overdose prevention, as well as resources such as naloxone, suicide hotlines, mental health, and substance use treatment. It will be available online and in print.
  Arms: Brief intervention (BI) then Enhanced Usual Care (EUC); Enhanced Usual Care (EUC) then EUC; Enhanced Usual Care (EUC) then Portal

SUMMARY:
The purpose of the study is to develop and test innovative interventions to prevent the development of opioid misuse and opioid use disorders among older adolescents and young adults (AYA; ages 16-30) who use opioids, which will be initiated from a health care visit in the emergency department and extended post discharge via a telehealth approach. This study will have significant impact by identifying optimal, cost-effective opioid prevention strategies to sustain outcomes among AYAs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-30 years
* Seeking care in Michigan Medicine emergency department (ED)
* Ability to read/comprehend and communicate in English
* Medically & cognitively able to provide consent or assent
* Prescription opioid use plus >=1 other risk factor (misuse positive for marijuana, other illicit drugs, other prescription drug misuse; binge drinking; depression or suicidality) or opioid misuse [prescription opioid misuse or illicit opioid use (e.g., heroin, fentanyl)]

Exclusion Criteria:

* Presenting with acute sexual assault, acute suicidality or a current cancer diagnosis/are currently receiving cancer treatment
* Current pregnancy at baseline
* History of injection drug use within last 12 months
* High risk for opioid use disorder
* Enrolled in Aim 1

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1155 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Change in opioid misuse | 3, 6, and 12 months
  Alcohol Smoking and Substance Involvement Screening Test severity score (prescription opioids/heroin, scores range 0-27 per subscale, higher score indicates worse outcomes)

SECONDARY OUTCOMES:
Change in days of opioid misuse | 3, 6, and 12 months
  Addiction Severity Index (modified; score ranges from 0-60, higher score indicates worse outcomes)
Change in overdose risk behaviors | 3, 6, and 12 months
  Opioid-related risk behaviors (score ranges from 0-32, higher score indicates worse outcomes)
Change in other drug and alcohol use | 3, 6, and 12 months
  Substance use index (based on frequency measures, higher scores indicate worse outcome)
Change in substance use consequences | 3, 6, and 12 months
  Adapted alcohol, cannabis, and/or opioid-related consequences (total, higher score indicates worse outcomes)
Change in impaired driving | 3, 6, and 12 months
  Adapted items from Young Adult Driving Questionnaire (5 items; score ranges from 0-30; higher score indicates worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Walton, PhD, Principal Investigator — University of Michigan; Erin Bonar, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuklinski MR, Gibbons BJ, Bowser DM, McCollister KE, Smart R, Dunlap LJ, Shenkar E, Bonar EE, Boomer T, Campbell M, Fiellin LE, Hutton DW, Rao V, Saldana L, Su K, Walton MA, Yilmazer T. Investing in Interventions to Prevent Opioid Use Disorder in Adolescents and Young Adults: Start-up Costs from NIDA's HEAL Prevention Initiative. Prev Sci. 2025 Nov;26(7):1045-1055. doi: 10.1007/s11121-025-01835-6. Epub 2025 Oct 14. PMID 41085955
- [Derived] Seewald L, Bonar E, Bohnert ASB, Carter PM, King CA, Losman ED, Bacon L, Wheeler T, Walton M. Lifetime non-fatal overdose experiences among at-risk adolescents and young adults in the emergency department with past-year opioid use in the USA. Inj Prev. 2024 Oct 1;30(5):373-380. doi: 10.1136/ip-2023-045072. PMID 38331586
- [Derived] Bonar EE, Kidwell KM, Bohnert ASB, Bourque CA, Carter PM, Clark SJ, Glantz MD, King CA, Losman ED, McCabe SE, Philyaw-Kotov ML, Prosser LA, Voepel-Lewis T, Zheng K, Walton MA. Optimizing scalable, technology-supported behavioral interventions to prevent opioid misuse among adolescents and young adults in the emergency department: A randomized controlled trial protocol. Contemp Clin Trials. 2021 Sep;108:106523. doi: 10.1016/j.cct.2021.106523. Epub 2021 Aug 2. PMID 34352386

DOCUMENTS (1):
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT04550715/ICF_000.pdf